CLINICAL TRIAL: NCT00905658
Title: Systematic Nutritional Care in Patients Receiving First-line Chemotherapy for Metastatic Gynecologic Cancer in a Phase II Study
Brief Title: Nutritional Supplements in Improving Quality of Life During First-Line Chemotherapy in Patients With Metastatic Gynecological Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000633553; COL-NUTRYS; COL-2007-06; COL-IDRCB-2007-A00454-49; INCA-RECF0634
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
Keywords: stage IVA cervical cancer; stage IVB cervical cancer; fallopian tube cancer; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; stage IV endometrial carcinoma; stage IV uterine sarcoma; stage IVA vaginal cancer; stage IVB vaginal cancer; stage IV vulvar cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial

ARMS (3):
- Arm I (No Intervention): Patients are monitored via standard follow-up assessments every 3 weeks.
  Interventions: Procedure: standard follow-up care
- Arm II (Experimental): Patients receive nutritional supplements and are monitored via standard follow-up assessments every 3 weeks.
  Interventions: Dietary Supplement: therapeutic nutritional supplementation; Procedure: standard follow-up care
- Arm III (Experimental): Patients receive nutritional supplements and are monitored via standard follow-up assessments every 3 weeks with additional biweekly assessments completed at home by a service provider.
  Interventions: Dietary Supplement: therapeutic nutritional supplementation; Procedure: standard follow-up care

INTERVENTIONS:
Dietary Supplement: therapeutic nutritional supplementation — Patients receive systematic nutritional supplementation
  Arms: Arm II; Arm III
Procedure: standard follow-up care — Patients undergo standard monitoring

SUMMARY:
RATIONALE: Learning about the effect of nutritional supplements on quality of life in patients receiving chemotherapy for cancer may help doctors plan the best treatment.

PURPOSE: This randomized phase II trial is studying nutritional supplements to see how well they work in improving quality of life during first-line chemotherapy in patients with metastatic gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Measure quality of life (QLQ-C30) at week 18 in patients with metastatic gynecological cancer receiving systematic nutritional supplements during first-line chemotherapy.

Secondary

* Study the maintenance or improvement of intake and nutritional status.
* Study the quality of life during chemotherapy.
* Evaluate tolerance and compliance to treatment with nutritional supplements.
* Evaluate the feasibility of and the tolerance to chemotherapy.
* Measure the overall survival over 18 weeks.
* Analyze the cost-effectiveness of different strategies of nutritional care.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients are monitored via standard follow-up assessments every 3 weeks.
* Arm II: Patients receive nutritional supplements and are monitored via standard follow-up assessments every 3 weeks.
* Arm III: Patients receive nutritional supplements and are monitored via standard follow-up assessments every 3 weeks with additional biweekly assessments completed at home by a service provider.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gynecological cancer

  * Currently receiving first-line chemotherapy for metastatic disease

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 or Karnofsky PS 70-100%
* Not pregnant or nursing
* Intake < 75% of theoretical need
* Weight loss ≥ 5% within the past 6 months
* No patients with dementia or altered mental status
* No psychological, familial, social, or geographic situations that preclude clinical follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent radiotherapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rodrigues-Lebrun, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France